CLINICAL TRIAL: NCT05063227
Title: Predictive Value of Different Nociception Monitoring Systems for the Prediction of Moderate to Severe Postoperative Pain After General Anesthesia
Brief Title: Prediction of Postoperative Pain by Nociception Monitoring
Acronym: PredictPain
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-06
Record Dates: First submitted 2021-07-10; First posted 2021-10-01 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Pain, Postoperative; Analgesia; Anesthesia Recovery Period; Opioid Use
Keywords: Analgesia Monitoring; General anesthesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Heart Rate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: As this is a single-group, observational study all patients will be monitored with all three nociception monitoring systems (the Surgical Pleth Index (SPI), the Pupillary Pain Index (PPI) and the Nociception Level (NOL)) and data on heart rate changes as a variable used in current clinical practice to choose the opioid dosage during general anesthesia will be obtained additionally.
  Interventions: Diagnostic Test: Observational: analgesia monitoring indices and changes in heart rate

INTERVENTIONS:
Diagnostic Test: Observational: analgesia monitoring indices and changes in heart rate — After the end of surgery (defined as the time of skin closure or wound dressing), but before awakening (BIS will still be < 60), SPI, PPI and NOL are recorded in a quiet setting without any other stimulation. Within the five minutes data acquisition period nociception indices are recorded every minute (T0, T1, T2, T3, T4, T5). The highest SPI, PPI and NOL are used for further analysis.

SUMMARY:
General anesthesia is a combination of hypnotic drugs and opioid analgesics. Modern general anesthesia aims to treat nociception induced by surgical stimulation while avoiding an overdose of opioid analgesics and reducing side-effects of opioid administration. Quality and safety of general anesthesia are of major clinical importance and can be improved by adjusting the opioid analgesics to the optimal individual dose needed. In the current clinical practice, the opioid dosage is usually chosen by clinical judgment, though recently different monitoring devices estimating the effect of nociception during unconsciousness have become commercially available. Nevertheless, the impact of nociception-monitor-guided opioid administration on the administered amount of opioid, postoperative short-term recovery, and long-term outcome is inconclusive. This study aims to investigate the predictive power of different nociception monitoring systems for the prediction of moderate to severe immediate postoperative pain from nociception indices measured before awakening from general anesthesia.

DETAILED DESCRIPTION:
General anesthesia is a combination of hypnotic drugs and opioid analgesics. Modern general anesthesia aims to treat nociception induced by surgical stimulation while avoiding an overdose of opioid analgesics and reducing side-effects of opioid administration. Underdosing of opioids during surgery can lead to nociception with increased sympathetic tone, elevated levels of stress hormones, unintended patient movement due to nociception as well as increased postoperative pain. On the other hand, overdosing of opioids can lead to negative side effects such as nausea and vomiting, arterial hypotension, immunosuppression, prolonged recovery times, postoperative delirium and an increase in postoperative pain by opioid-induced-hyperalgesia. Quality and safety of general anesthesia are of major clinical importance and can be improved by adjusting the opioid analgesics to the optimal individual dose needed. In the current clinical practice, the opioid dosage is chosen by clinical judgment of the attending anesthesiologist based on changes in the heart rate, blood pressure, pupil size, lacrimation and sweating of the patient. In recent years, different monitoring devices estimating the effect of nociception during unconsciousness have become commercially available. These monitoring devices use several different mechanisms, such as heart rate (HR) variability, pulse wave photoplethysmography, pupil reflex dilation, and skin conductance measurement, and based on these signals index the nociception/analgesia balance. Such monitoring devices should help physicians choose the right dose of opioid analgesics during general anesthesia. Nevertheless, the impact of nociception-monitor-guided opioid administration on the administered amount of opioid, postoperative short-term recovery, and long-term outcome is inconclusive.

Current literature is inconclusive if the nociception monitoring devices have predictive power to predict immediate postoperative pain after awakening from general anesthesia already before awakening from general anesthesia.

In this prospective, double-blinded, observational clinical study the investigators aim to evaluate the predictive power of different nociception monitoring systems for the prediction of moderate to severe immediate postoperative pain from nociception indices measured before awakening from general anesthesia. The nociception monitoring systems included in the study are the Surgical Pleth Index (SPI), the Pupillary Pain Index (PPI) and the Nociception Level (NOL) and heart rate changes as a variable used in current clinical practice to choose the opioid dosage during general anesthesia.

The postoperative pain level will be assessed from anesthesia nurses using the Numerical Rating Scale (NRS) who are blinded to the nociception indices measured before awakening.

For SPI monitoring there are findings suggesting that an SPI > 30 could be the 'best-fit' optimal threshold with the highest sum of sensitivity and specificity to detect moderate to severe pain. Nevertheless, positive and negative predictive value of SPI were still rather low.

For PPI monitoring there are data demonstrating a moderate correlation between PPI values before tracheal extubation and postoperative pain. Another study with pupil dilatation reflex threshold showed only a minor correlation between pupil dilatation reflex threshold and the intensity of immediate postoperative pain.

For NOL monitoring, on the one hand, there are data suggesting that a threshold of > 20 after knife to skin incision has predictive power to predict moderate to severe postoperative pain. On the other hand, the highest combined sensitivity and specificity were still rather low. While a NOL < 10 after skin incision excluded moderate-severe postoperative pain with a negative predictive value of 83%, the NOL during surgery and at the end of surgery did not allow the exclusion or the prediction of moderate-severe postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with elective trauma surgery and orthopedic surgery scheduled on a weekday Monday to Friday in the operation theater where the study is conducted

Exclusion Criteria:

* Beta blocker, digitalis or cardiac pacemaker therapy
* Higher degrees of cardiac arrhythmias, e.g. atrial fibrillation and atrio-ventricular block >1st degree
* Severe peripheral or cardiac neuropathy
* Eye disease with affection of pupil reactivity
* Intraoperative treatment with ketamine, beta-receptor blockers, beta-receptor agonists or clonidine and treatment with vasoactive medication within 10 min before and during data acquisition period
* Inability to adequately specify postoperative pain level
* Postoperative care in the intensive care unit (ICU) or postanesthesia care unit with planned overnight stay (PACU24, intermediate care unit IMC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes all patients with elective trauma surgery and orthopedic surgery scheduled on a weekday Monday to Friday in the operation theater where the study is conducted,which do not present with an exclusion criterion. There is no further eligibility criteria and thusly, this is a non-sepcified study on all patients that meet the requirements for the three analgesia monitoring devices.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Primary endpoint will be the diagnostic accuracy (ROC analysis) of the nociception indices after the end of surgery to predict moderate to severe immediate postoperative pain | Once immediately after arrival in the post-anesthesia care unit (PACU)
  Numerical Rating Scale (NRS) Scale 4-10 NRS has a minimal value of 0 and a maximal value of 10, higher scores mean a worse outcome (higher pain level).

SECONDARY OUTCOMES:
The correlation between the nociception indices after the end of surgery and immediate postoperative pain measured with the NRS on a scale of 0 - 10 | Once immediately after arrival in the post-anesthesia care unit (PACU)
  Numerical Rating Scale (NRS) NRS has a minimal value of 0 and a maximal value of 10, higher scores mean a worse outcome (higher pain level).
The correlation between the nociception indices after the end of surgery and postoperative pain measured with the NRS on a scale of 0 - 10 after 60 minutes in PACU | First 60 minutes after arrival in the PACU
  Numerical Rating Scale (NRS) NRS has a minimal value of 0 and a maximal value of 10, higher scores mean a worse outcome (higher pain level).
Correlation between the nociception indices and the highest postoperative NRS | Once in the first 2 hours during the PACU stay
  Numerical Rating Scale (NRS) NRS has a minimal value of 0 and a maximal value of 10, higher scores mean a worse outcome (higher pain level).
The correlation between the nociception indices after the end of surgery and the amount of opioids in the first 30 minutes after surgery | Time period of first 30 minutes during the PACU stay
  Cumulative amount of opioids in morphine equivalents
The correlation between the nociception indices after the end of surgery and the amount of opioids in up to 2 hours after surgery | Time period of first 2 hours during the PACU stay
  Cumulative amount of opioids in morphine equivalents

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Nitzschke, MD, Principal Investigator — Center for Anesthesiology and Intensive Care Medicine, University Medical Center Hamburg-Eppendorf
Locations (1):
- Rainer Nitzschke, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data on request only.

REFERENCES:
- [Derived] Koschmieder KC, Funcke S, Shadloo M, Pinnschmidt HO, Greiwe G, Fischer M, Nitzschke R. Validation of three nociception indices to predict immediate postoperative pain before emergence from general anaesthesia: a prospective double-blind, observational study. Br J Anaesth. 2023 Apr;130(4):477-484. doi: 10.1016/j.bja.2022.11.024. Epub 2023 Jan 4. PMID 36609057